CLINICAL TRIAL: NCT02658604
Title: Home Medication Review Services for Non-homebound Community Pharmacy Patients: Evaluation of Medication Management Issues in Non-homebound Patients and Characterization of Ideal Target Population for Home-based Medication Reviews.
Brief Title: Home Medication Reviews by Pharmacists in Ontario, Canada
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Sherilyn Houle, Assistant Professor, University of Waterloo
Other Study IDs: 20836
Record Dates: First submitted 2016-01-13; First posted 2016-01-20 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Home Care; Pharmacists; Medication Therapy Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Home visit by pharmacist: Patients of participating pharmacies age 65 or older, who are on 5 or more chronic prescription medications, and who have a need for, and agree to, a home visit by a pharmacist for a medication review.
  Interventions: Other: Home medication review by a pharmacist

INTERVENTIONS:
Other: Home medication review by a pharmacist — Patients will receive a home visit from a pharmacist, including a medication review and the identification and addressing of drug therapy problems through patient education, the provision of pharmacologic and/or non-pharmacologic advice, or the adaptation of therapy or communication of recommendations to prescribers. All activities are within the current scope of practice for pharmacists in Ontario. A detailed assessment of the patient's medication inventory and organization/storage practices will be conducted, followed by a medication cabinet cleanup to help the patient organize their medications and discard any expired or discontinued medications. A list of inappropriate medications found in the home will be documented, detailing the reasons why they are inappropriate and if/how the patient is currently using these medications. With patient consent, inappropriate medications will be removed from the home and returned to the pharmacy for safe disposal.

SUMMARY:
RATIONALE:

Several examples in the literature describe the types of medication management issues uncovered during the course of home-based medication reviews. For example, the investigators previously reported the outcomes of home medication reviews of 43 homebound community pharmacy patients, finding that 58% of patients were keeping medications in the home that were expired, duplicates of other current medications, or no longer therapeutically appropriate.

Many of these issues, due to their nature, could be considered to be "hidden", i.e. issues that are unlikely to be adequately detected or resolved during the course of routine interactions between patients and pharmacists in the community pharmacy setting. Currently, only homebound patients in Ontario are eligible to receive government-funded home medication review services from pharmacists. This limitation in funding eligibility is problematic as it reduces the likelihood that non-homebound patients will receive home medication reviews, even though this population may also benefit from these services. Indeed, evidence in the literature is not limited exclusively to homebound patients, and suggests that non-homebound patients are also at risk from home-centered medication management issues and may also benefit from home medication reviews.

PURPOSE:

Our study aims to characterize the prevalence and nature of "hidden in the home" medication management issues in non-homebound patients. To our knowledge, this study would be the first of its kind to focus specifically on this patient population and lend direct evidence in support of expanding funding of home medication review services in Ontario to include non-homebound patients.

HYPOTHESIS:

A subset of ambulatory, non-homebound patients who regularly attend community pharmacies are affected by medication management issues that cannot be adequately identified and resolved during the course of a typical medication review taking place within the pharmacy. These patients would benefit from a full medication review taking place in their own homes, similar to what is presently provided under Ontario's MedsCheck at Home program, for which only homebound patients in Ontario are eligible.

RESEARCH QUESTIONS/OBJECTIVES:

1. What is the frequency of, and what type(s) and severity of, drug-related problems are detected during pharmacist visits to patients' homes who would not otherwise qualify for a MedsCheck at Home service?
2. Based on the findings from this study, which criteria would best assist community pharmacists in identifying ambulatory patients who may stand to benefit most from a home-based medication review?

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* On 5 or more chronic prescription medications
* Score of 3/8 or higher on screening questionnaire
* Live at home and are ambulatory
* Willingness to have a pharmacist conduct a medication review in their home

Exclusion Criteria:

* Unable to converse with the pharmacist in a language they both can communicate in

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Current patients of participating pharmacies who are aged 65 and older, live at home, and are on 5 or more medications.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Mean number of drug therapy problems (DTP) identified per patient | At time of home visit (cross-section), up to 6 months
  DTP definitions based on those of Hepler and Strand (1990)

SECONDARY OUTCOMES:
Frequency distribution of drug therapy problem (DTP) type(s) across patient population | At time of home visit (cross-section), up to 6 months
  DTP definitions based on those of Hepler and Strand (1990)

OTHER OUTCOMES:
Mean number of high-risk medications used per patient | At time of home visit (cross-section), up to 6 months
  High-risk medications are those defined by the Beers' Criteria

CONTACTS AND LOCATIONS:
Overall Officials: John Papastergiou, BSc, BScPhm, Principal Investigator — University of Waterloo
Locations (1):
- Shoppers Drug Mart #500, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No